CLINICAL TRIAL: NCT07103655
Title: The Therapeutic Value of Mavacamten in Hypertrophic Cardiomyopathy With Mid-to-Apical Left Ventricular Obstruction: A Prospective, Interventional, Real-World Clinical Study.
Brief Title: The Therapeutic Value of Mavacamten in Hypertrophic Cardiomyopathy With Mid-to-Apical Left Ventricular Obstruction
Acronym: BRAVE-HCM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, xie xiaojie, MD, PhD, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1056
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461; Adrenergic beta-Antagonists; Metoprolol; Bisoprolol; Carvedilol; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mavacamten (Experimental): Add-on use of mavacamten on top of guideline-directed standard medical therapy
  Interventions: Drug: mavacamten; Drug: Beta Blocker (BB) - metoprolol, bisoprolol, carvedilol; Drug: diltiazem
- No mavacamten (Active Comparator): Guideline-directed standard medical therapy group
  Interventions: Drug: Beta Blocker (BB) - metoprolol, bisoprolol, carvedilol; Drug: diltiazem

INTERVENTIONS:
Drug: mavacamten — Add Mavacamten to guideline-directed standard medical therapy for patients with hypertrophic cardiomyopathy (HCM) and mid-to-apical left ventricular obstruction.
  Other Names: beta receptor blockers
  Arms: Mavacamten
Drug: Beta Blocker (BB) - metoprolol, bisoprolol, carvedilol — Administer an appropriate dose of beta-blockers according to the patient's tolerance.
Drug: diltiazem — Administer an appropriate dose of diltiazem according to the patient's tolerance.

SUMMARY:
This study is a prospective interventional cohort study aimed at evaluating the therapeutic efficacy and clinical utility of Mavacamten-a targeted myosin inhibitor specifically developed for obstructive hypertrophic cardiomyopathy (HCM)-in patients with HCM characterized by mid-to-apical left ventricular obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HCM according to the 2023 Chinese Guidelines for the Diagnosis and Treatment of Adult Hypertrophic Cardiomyopathy, meeting one of the following:

  1. Left ventricular wall thickness ≥15 mm at end-diastole in any segment as assessed by echocardiography or cardiac magnetic resonance imaging (CMR);
  2. Left ventricular wall thickness ≥13 mm in individuals with a confirmed pathogenic gene mutation or in genetically affected family members;
  3. Exclusion of other cardiovascular, systemic, or metabolic disorders that may cause ventricular hypertrophy.

     * Symptomatic non-outflow tract obstructive HCM patients (meeting criterion a and at least one of b or c):

  <!-- -->

  1. Presence of clinical symptoms such as dyspnea, chest pain, dizziness, palpitations, or syncope, with New York Heart Association (NYHA) functional class II-III;
  2. Maximal pressure gradient (PGmax) >30 mmHg in the mid-ventricle under resting or Valsalva maneuver as assessed by echocardiography;
  3. PGmax >30 mmHg in the apical region under resting or Valsalva maneuver on echocardiography.

     ③Ability to provide written informed consent (ICF) and any required privacy authorization prior to study enrollment.

     Exclusion Criteria:

     -
* Obstructive hypertrophic cardiomyopathy (HCM), defined as a maximal left ventricular outflow tract pressure gradient (LVOT-PGmax) ≥30 mmHg at rest and during the Valsalva maneuver on echocardiography;

  * Maximal right ventricular outflow tract pressure gradient (RVOT-PGmax) ≥16 mmHg at rest; ③ Left ventricular ejection fraction (LVEF) <50% on echocardiography;

    * Uncontrolled primary hypertension;

      * Moderate or severe aortic valve stenosis and/or primary mitral valve disease with severe mitral regurgitation; ⑥ Known infiltrative or storage disorders mimicking the HCM phenotype (e.g., Fabry disease, cardiac amyloidosis); ⑦ Presence of severe infections, hepatic dysfunction, renal impairment, or other serious conditions significantly affecting life expectancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage change in pressure gradient during the Valsalva maneuver | Week 36
  The percentage reduction in the pressure gradient at the site of left ventricular obstruction during the Valsalva maneuver at week 36, compared to baseline, as measured by echocardiography.

SECONDARY OUTCOMES:
Anterior papillary muscle to the interventricular septum distance | Week 36
  Percentage Increase in the distance from the anterior papillary muscle to the interventricular septum
Left atrial global longitudinal strain | Week 36
  Left Atrial Global Longitudinal Strain (LA GLS) is an echocardiographic parameter derived from speckle-tracking imaging that measures the longitudinal deformation of the left atrial myocardium throughout the cardiac cycle.
Left ventricular global longitudinal strain | Week 36
  Left Ventricular Global Longitudinal Strain (LVGLS) is a sensitive echocardiographic parameter derived from speckle-tracking imaging that quantifies the myocardial deformation in the longitudinal direction. It reflects the shortening of myocardial fibers along the long axis of the left ventricle during systole.
Percentage change in resting pressure gradient | Week 36
  The percentage reduction in the pressure gradient at the site of left ventricular obstruction at rest measured by echocardiography at week 36 compared to baseline.
Absolute change in pressure gradient during the Valsalva maneuver | Week 36
  The absolute decrease in number of the pressure gradient at the site of left ventricular obstruction during the Valsalva maneuver measured by echocardiography at week 36 compared to baseline.
The proportion of patients with a pressure gradient <30 mmHg during the Valsalva maneuver | Week 36
  The proportion of patients with a pressure gradient <30 mmHg at the site of obstruction during the Valsalva maneuver at week 36.
BNP | Week 36
  Number decrease in BNP levels from baseline to week 36.
Troponin T | Week 36
  Number decrease in Troponin T levels from baseline to week 36.
New-onset atrial fibrillation | From baseline to week 36
  Rate of new-onset atrial fibrillation in each group during the study period
LVEF<50% | From baseline to week 36
  The proportion of patients in each group with LVEF <50% accompanied by signs and symptoms of heart failure worsening and/or an increase in BNP of ≥30% compared to the previous measurement during the study period.
LVEF<40% | From baseline to week 36
  Rate of LVEF <40% in each group during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided